CLINICAL TRIAL: NCT02487810
Title: Intuition Versus Deliberation in Decisions About Life-Sustaining Medical Therapies
Brief Title: Intuition vs. Deliberation in Medical Decision Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Leonard Davis Institute (Unknown)
Responsible Party: Principal Investigator, Scott Halpern, Assistant Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UPenn 822238
Record Dates: First submitted 2015-06-25; First posted 2015-07-02 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-05

CONDITIONS: Decision Making About Life-sustaining Treatment in Patients With Serious Cardiac, Respiratory and Oncological Conditions Likely to Limit Life Expectancy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intuitive (Experimental): Patients in each arm will be asked all of the same questions. The only difference between the arms will be the instructions regarding how and when to answer the series of hypothetical questions regarding medical interventions. The instructions will be designed to influence patients to think either intuitively or deliberatively about the questions regarding life-sustaining interventions.
  Interventions: Behavioral: Cognitive load
- Deliberative (Experimental): Patients in each arm will be asked all of the same questions. The only difference between the arms will be the instructions regarding how and when to answer the series of hypothetical questions regarding medical interventions. The instructions will be designed to influence patients to think either intuitively or deliberatively about the questions regarding life-sustaining interventions.
  Interventions: Behavioral: Deliberative instructions

INTERVENTIONS:
Behavioral: Cognitive load — Patients in the intuition arm of the study will be asked to complete a memorization task while they are answering survey questions.
  Arms: Intuitive
Behavioral: Deliberative instructions — Patients in the deliberative arm will be given instructions to take their time and deliberate on their decisions
  Arms: Deliberative

SUMMARY:
The purpose of this study is to determine whether there are systematic differences between the decisions patients make intuitively versus deliberatively about life-sustaining medical therapies.

The targeted population is inpatients at the Hospital of the University of Pennsylvania with serious medical problems. The study will involve facilitated interviews with patients using a survey instrument developed in Qualtrics.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 and older
2. Currently an inpatient at Hospital of the University of Pennsylvania
3. Speaks and reads fluently in English
4. Either

   1. Has one of the following medical conditions:

      * Chronic obstructive pulmonary disease with at least severe airflow obstruction on most recent spirometry and/or eligible for long-term oxygen therapy
      * Incurable interstitial lung disease with at least severe restriction on most recent pulmonary function tests and/or eligible for long-term oxygen therapy
      * Congestive heart failure with NYHA Class III or higher and current hospitalization related to heart failure
      * Acute myeloid leukemia
      * Stage IV lymphoma
      * Stage IIIB or Stage IV non-small cell lung cancer, cholangiocarcinoma, renal cell carcinoma, breast cancer, uterine cancer, cervical cancer, ovarian cancer, colorectal cancer, gastric cancer, pancreatic cancer, prostate cancer, urothelial cancer
      * Stage C or D hepatocellular carcinoma
      * Mesothelioma or any malignancy metastatic to the pleura; or
   2. Is hospitalized on oncology, pulmonary or cardiology service and has been hospitalized at least one other time during the last year on the same service
5. Stable vital signs

Exclusion Criteria:

1. Notation of code status limitation in electronic medical record
2. Cognitive impairment to the point unable to give informed consent
3. Current feeding tube placement
4. Current tracheostomy
5. Severe pain, shortness of breath or other uncontrolled symptoms
6. Actively undergoing evaluation for solid organ transplant
7. First hospitalization after diagnosis of serious illness

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Halpern, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Rubin EB, Buehler AE, Cooney E, Gabler NB, Mante AA, Halpern SD. Intuitive vs Deliberative Approaches to Making Decisions About Life Support: A Randomized Clinical Trial. JAMA Netw Open. 2019 Jan 4;2(1):e187851. doi: 10.1001/jamanetworkopen.2018.7851. PMID 30681717

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intuitive | Deliberative
Started | 98 | 102
Completed | 97 | 102
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intuitive | Deliberative | Total
Number analyzed (Participants) | 97 | 102 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (4.8) | 67.9 (5.2) | 67.2 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 67
  Male | 64 | 68 | 132

OUTCOME MEASURES:

1. Primary Outcome: Acceptance or Refusal of a Feeding Tube for Chronic Aspiration
Description: Patients in each arm will be asked all of the same questions. The only difference between the arms will be the instructions regarding how and when to answer the series of hypothetical questions regarding acceptance of a feeding tube for chronic aspiration. In this hypothetical scenario, patients are presented with a situation in which they are unable to eat or drink safely such that small amounts of food or liquid go to their lungs and cause trouble with breathing. The instructions will be designed to influence patients to think either intuitively or deliberatively about the questions regarding life-sustaining interventions. Cognitive load: Patients in the intuition arm of the study will be asked to complete a memorization task while they are answering survey questions.
Time Frame: The trial involves a questionnaire that will be given on a single day; patients will not be followed longitudinally
Measure: Count of Participants; unit: Participants
Arm/Group | Intuitive Arm | Deliberative Arm
Number analyzed (Participants) | 97 | 102
Participants
  Accept Feeding Tube | 41 | 45
  Reject Feeding Tube | 56 | 57

2. Primary Outcome: Acceptance or Refusal of Antibiotics
Description: Patients in each arm will be asked all of the same questions. The only difference between the arms will be the instructions regarding how and when to answer the series of hypothetical questions regarding acceptance of antibiotics. In this hypothetical scenario, patients are presented with an illness severity such that they drift in and out of consciousness some days and are expected to die in several months. The instructions will be designed to influence patients to think either intuitively or deliberatively about the questions regarding life-sustaining interventions. Cognitive load: Patients in the intuition arm of the study will be asked to complete a memorization task while they are answering survey questions.
Time Frame: The trial involves a questionnaire that will be given on a single day; patients will not be followed longitudinally
Measure: Count of Participants; unit: Participants
Arm/Group | Intuitive Arm | Deliberative Arm
Number analyzed (Participants) | 97 | 102
Participants
  Accept antibiotics | 38 | 44
  Refuse antibiotics | 59 | 58

3. Primary Outcome: Acceptance or Refusal of Breathing Machine
Description: Patients in each arm will be asked all of the same questions. The only difference between the arms will be the instructions regarding how and when to answer the series of hypothetical questions regarding acceptance of a breathing machine. In this hypothetical scenario, patients are presented with a life-threatening illness with 50% chance of survival provided that they receive support from a breathing machine for two weeks. The instructions will be designed to influence patients to think either intuitively or deliberatively about the questions regarding life-sustaining interventions. Cognitive load: Patients in the intuition arm of the study will be asked to complete a memorization task while they are answering survey questions.
Time Frame: The trial involves a questionnaire that will be given on a single day; patients will not be followed longitudinally
Measure: Count of Participants; unit: Participants
Arm/Group | Intuitive Arm | Deliberative Arm
Number analyzed (Participants) | 97 | 102
Participants
  Accept intubation | 57 | 61
  Refuse intubation | 40 | 41

4. Primary Outcome: Acceptance or Refusal of Tracheostomy
Description: Patients in each arm will be asked all of the same questions. The only difference between the arms will be the instructions regarding how and when to answer the series of hypothetical questions regarding acceptance of a tracheostomy and support from a breathing machine for at least two months to survive. The instructions will be designed to influence patients to think either intuitively or deliberatively about the questions regarding life-sustaining interventions. Cognitive load: Patients in the intuition arm of the study will be asked to complete a memorization task while they are answering survey questions.
Time Frame: The trial involves a questionnaire that will be given on a single day; patients will not be followed longitudinally
Measure: Count of Participants; unit: Participants
Arm/Group | Intuitive Arm | Deliberative Arm
Number analyzed (Participants) | 97 | 102
Participants
  Accept tracheostomy | 36 | 42
  Refuse tracheostomy | 61 | 60

5. Secondary Outcome: Scores on Uncertainty Subscale of Decisional Conflict Scale
Description: Decisional uncertainty will be evaluated using the uncertainty subscale of the Decisional Conflict Scale ranging from 0-100 such that 0 = extremely CERTAIN about best choice and 100 = extremely UNCERTAIN about the best choice. Higher values represent MORE UNCERTAINTY with decisions regarding feeding tubes, antibiotics, intubation, and tracheostomy while lower values represent LESS UNCERTAINTY.
Time Frame: The trial involves a questionnaire that will be given on a single day; patients will not be followed longitudinally
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intuitive Arm | Deliberative Arm
Number analyzed (Participants) | 97 | 102
units on a scale
  Feeding Tube | 21.5 (23.1) | 20.9 (21.1)
  Antibiotics | 20.3 (21.7) | 18.9 (21.2)
  Intubation | 26.2 (25.5) | 20.8 (22.1)
  Tracheostomy | 29.4 (25.3) | 23.6 (24.8)

6. Secondary Outcome: Correlation Between Accepting Tracheostomy and Thinking That Being Bed Bound is Equal to or Worse Than Death
Description: This outcome measures the proportion of participants who accept tracheostomy AND indicate that bed bound is a state that is either equal to, or worse than death. This proportion will be measured separately in the deliberative and intuitive groups; these proportions will then be compared.
Time Frame: The trial involves a questionnaire that will be given on a single day; patients will not be followed longitudinally
Measure: Count of Participants; unit: Participants
Arm/Group | Intuitive Arm | Deliberative Arm
Number analyzed (Participants) | 26 | 37
Participants
  Accept tracheostomy | 4 | 9
  Refuse tracheostomy | 22 | 28

7. Secondary Outcome: Correlation Between Accepting Antibiotics and Thinking That Being Bed Bound is Equal to or Worse Than Death.
Description: This outcome measures the proportion of participants who accept antibiotics AND indicate that bed bound is a state that is either equal to, or worse than death. This proportion will be measured separately in the deliberative and intuitive groups; these proportions will then be compared.
Time Frame: The trial involves a questionnaire that will be given on a single day; patients will not be followed longitudinally
Measure: Count of Participants; unit: Participants
Arm/Group | Intuitive Arm | Deliberative Arm
Number analyzed (Participants) | 26 | 37
Participants
  Accept Antibiotics | 6 | 13
  Refuse Antibiotics | 20 | 24

8. Secondary Outcome: Correlation Between Accepting Tracheostomy and Thinking That Needing Care All the Time is Equal to or Worse Than Death
Description: This outcome measures the proportion of participants who accept tracheostomy AND indicate that needing care all the time is a state that is either equal to, or worse than death. This proportion will be measured separately in the deliberative and intuitive groups; these proportions will then be compared.
Time Frame: The trial involves a questionnaire that will be given on a single day; patients will not be followed longitudinally
Measure: Count of Participants; unit: Participants
Arm/Group | Intuitive Arm | Deliberative Arm
Number analyzed (Participants) | 21 | 25
Participants
  Accept Tracheostomy | 2 | 8
  Refuse Tracheostomy | 19 | 17

9. Secondary Outcome: Correlation Between Accepting Antibiotics and Thinking That Needing Care All the Time is Equal to or Worse Than Death
Description: This outcome measures the proportion of participants who accept antibiotics AND indicate that needing care all the time is a state that is either equal to, or worse than death. This proportion will be measured separately in the deliberative and intuitive groups; these proportions will then be compared.
Time Frame: The trial involves a questionnaire that will be given on a single day; patients will not be followed longitudinally
Measure: Count of Participants; unit: Participants
Arm/Group | Intuitive Arm | Deliberative Arm
Number analyzed (Participants) | 21 | 25
Participants
  Accept Antibiotics | 4 | 9
  Refuse Antibiotics | 17 | 16

10. Secondary Outcome: Correlation Between Accepting Tracheostomy and Thinking That Living in a Nursing Home is Equal to or Worse Than Death
Description: This outcome measures the proportion of participants who accept tracheostomy AND indicate that living in a nursing home is a state that is either equal to, or worse than death. This proportion will be measured separately in the deliberative and intuitive groups; these proportions will then be compared.
Time Frame: The trial involves a questionnaire that will be given on a single day; patients will not be followed longitudinally
Measure: Count of Participants; unit: Participants
Arm/Group | Intuitive Arm | Deliberative Arm
Number analyzed (Participants) | 18 | 26
Participants
  Accept Tracheostomy | 4 | 5
  Refuse Tracheostomy | 14 | 21

11. Secondary Outcome: Correlation Between Accepting Antibiotics and Thinking That Living in a Nursing Home is Equal to or Worse Than Death
Description: This outcome measures the proportion of participants who accept antibiotics AND indicate that living in a nursing home is a state that is either equal to, or worse than death. This proportion will be measured separately in the deliberative and intuitive groups; these proportions will then be compared.
Time Frame: The trial involves a questionnaire that will be given on a single day; patients will not be followed longitudinally
Measure: Count of Participants; unit: Participants
Arm/Group | Intuitive Arm | Deliberative Arm
Number analyzed (Participants) | 18 | 26
Participants
  Accept Antibiotics | 5 | 8
  Refuse Antibiotics | 13 | 18

12. Secondary Outcome: Correlation Between Accepting Tracheostomy and Thinking That Relying on a Breathing Machine is Equal to or Worse Than Death
Description: This outcome measures the proportion of participants who accept tracheostomy AND indicate that relying on a breathing machine is a state that is either equal to, or worse than death. This proportion will be measured separately in the deliberative and intuitive groups; these proportions will then be compared.
Time Frame: The trial involves a questionnaire that will be given on a single day; patients will not be followed longitudinally
Measure: Count of Participants; unit: Participants
Arm/Group | Intuitive Arm | Deliberative Arm
Number analyzed (Participants) | 25 | 32
Participants
  Accept Tracheostomy | 4 | 7
  Refuse Tracheostomy | 21 | 25

13. Secondary Outcome: Correlation Between Accepting a Feeding Tube and Thinking That Relying on a Feeding Tube is Equal to or Worse Than Death
Description: This outcome measures the proportion of participants who accept a feeding tube AND indicate that relying on a feeding tube is a state that is either equal to, or worse than death. This proportion will be measured separately in the deliberative and intuitive groups; these proportions will then be compared.
Time Frame: The trial involves a questionnaire that will be given on a single day; patients will not be followed longitudinally
Measure: Count of Participants; unit: Participants
Arm/Group | Intuitive Arm | Deliberative Arm
Number analyzed (Participants) | 46 | 54
Participants
  Accept feeding tube | 7 | 16
  Refuse feeding tube | 39 | 38

ADVERSE EVENTS:
Description: This is a minimal risk study. We did not monitor for serious adverse events because 0 participants were at risk.
Arm/Group | Intuitive | Deliberative
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/97 | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No